CLINICAL TRIAL: NCT00797797
Title: A Multicenter, Randomized, Open-Label, Controlled Study to Evaluate the Safety, Tolerability, and Efficacy of Milnacipran When Added to Pregabalin in the Treatment of Fibromyalgia
Brief Title: Study of Milnacipran Added to Pregabalin for Treatment of Fibromyalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: James Perhach, Executive Director, Clinical Development, Forest Research Institute Inc (A Subsidiary of Forest Laboratories Inc)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MLN-MD-15
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Results first posted 2011-02-16 (Estimated); Last update posted 2011-02-16 (Estimated); Status verified 2011-01

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; milnacipran; pregabalin; treatment; Forest Research Institute
MeSH Terms: conditions — Fibromyalgia | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Milnacipran Added (Experimental)
  Interventions: Drug: Milnacipran Added
- No Treatment Added (Experimental)
  Interventions: Drug: No Treatment Added

INTERVENTIONS:
Drug: No Treatment Added — No added treatment
  Other Names: Lyrica (r)
  Arms: No Treatment Added
Drug: Milnacipran Added — Milnacipran 100 mg/d added
  Arms: Milnacipran Added

SUMMARY:
To evaluate the safety, tolerability, and efficacy of milnacipran when taken with another drug called pregabalin in people with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of fibromyalgia defined by 1990 American College of Rheumatology (ACR) Criteria
* tolerate at least 300 mg/day of pregabalin
* have an incomplete response to pregabalin treatment

Exclusion Criteria:

* suicidal risk
* substance abuse
* pulmonary dysfunction
* renal impairment
* active cardiac disease
* liver disease
* narrow angle glaucoma
* autoimmune disease
* cancer
* inflammatory bowel disease
* unstable endocrine disease
* prostatic enlargement

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2008-11; Primary Completion 2009-11 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia D'Astoli, Study Director — Forest Research Institute, a subsidiary of Forest Laboratories, Inc.
Locations (56):
- United States (56):
  - Forest Investigative Site, Birmingham, Alabama
  - Forest Investigative Site, Mesa, Arizona
  - Forest Investigative Site, Peoria, Arizona
  - Forest Investigative Site, Hot Springs, Arkansas
  - Forest Investigative Site, Anaheim, California
  - Forest Investigative Site, Sacramento, California
  - Forest Investigative Site, Torrance, California
  - Forest Investigative Site, Walnut Creek, California
  - Forest Investigative Site, Denver, Colorado
  - Forest Investigative Site, Cromwell, Connecticut
  - Forest Investigative Site, Danbury, Connecticut
  - Forest Investigative Site, Clearwater, Florida
  - Forest Investigative Site, Daytona Beach, Florida
  - Forest Investigative Site, Delray Beach, Florida
  - Forest Investigative Site, Fort Myers, Florida
  - Forest Investigative Site, Jacksonville, Florida
  - Forest Investigative Site, Miami, Florida
  - Forest Investigative Site, Ocala, Florida
  - Forest Investigative Site Orl2, Orlando, Florida
  - Forest Investigative Site, Orlando, Florida
  - Forest Investigative Site, Ormond Beach, Florida
  - Forest Investigative Site PP1, Pembroke Pines, Florida
  - Forest Investigative Site PP2, Pembroke Pines, Florida
  - Forest Investigative Site, Pismo Beach, Florida
  - Forest Investigative Site, St. Petersburg, Florida
  - Forest Investigative Site, Tampa, Florida
  - Forest Investigative Site, Atlanta, Georgia
  - Forest Investigative Site, Honolulu, Hawaii
  - Forest Investigative Site, Couer D'Alene, Idaho
  - Forest Investigative Site, Evansville, Indiana
  - Forest Investigative Site, Indianapolis, Indiana
  - Forest Investigative Site, Baltimore, Maryland
  - Forest Investigative Site, No. Dartmouth, Massachusetts
  - Forest Investigative Site, Worcester, Massachusetts
  - Forest Investigative Site, Jackson, Mississippi
  - Forest Investigative Site, St Louis, Missouri
  - Forest Investigative Site, Omaha, Nebraska
  - Forest Investigative Site, Albuquerque, New Mexico
  - Forest Investigative Site, Syracuse, New York
  - Forest Investigative Site, Cincinnati, Ohio
  - Forest Investigative Site, Cleveland, Ohio
  - Forest Investigative Site, Eugene, Oregon
  - Forest Investigative Site, Medford, Oregon
  - Forest Investigative Site, Portland, Oregon
  - Forest Investigative Site, Greer, South Carolina
  - Forest Investigative Site, Memphis, Tennessee
  - Forest Investigative Site, Houston, Texas
  - Forest Investigative Site, Lake Jackson, Texas
  - Forest Investigative Site, Salt Lake City, Utah
  - Forest Investigative Site, Woodstock, Vermont
  - Forest Investigative Site, Bellevue, Washington
  - Forest Investigative Site, Bellingham, Washington
  - Forest Investigative Site SEA1, Seattle, Washington
  - Forest Investigative Site SEA2, Seattle, Washington
  - Forest Investigative Site, Spokane, Washington
  - Forest Investigative Site, Racine, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and enrolled in this study within the US from December 2008 to June 2009.
Pre-assignment Details: Participants entered an open label pregabalin period concurrent with prohibited medication washout. Incomplete responders to pregabalin were randomized to receive either milnacipran (100 mg/d) or no added treatment for 11 weeks. All participant continued background stable dose pregabalin (300 or 450 mg/d) throughout the randomized treatment period.
Groups:
- No Treatment Added: No treatment added for 11 weeks of randomized treatment period
- Milnacipran Added: Milnacipran (100 mg/day) added for 11 weeks of randomized treatment period
Period: Overall Study
Arm/Group | No Treatment Added | Milnacipran Added
Started | 178 (Two patients took no background stable dose of pregabalin after randomization and are not included.) | 184
Completed | 123 | 141
Not Completed | 55 | 43

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Treatment Added | Milnacipran Added | Total
Number analyzed (Participants) | 178 | 184 | 362
Age Categorical [Number; unit: participants]
  Between 18 and 60 years | 151 | 146 | 297
  >=60 years | 27 | 38 | 65
Age Continuous [Mean (Standard Deviation); unit: years] | 48.8 (10.4) | 49.8 (10.3) | 49.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 170 | 329
  Male | 19 | 14 | 33
Region of Enrollment [Number; unit: participants]
  United States | 178 | 184 | 362

OUTCOME MEASURES:

1. Primary Outcome: Patient Global Impression of Change (PGIC) Responder Rate at End of Study
Description: The primary efficacy parameter was the PGIC responder rate, defined as the percentage of patients who rated themselves as "very much improved" or "much improved" (ie, having a score of 1 or 2 on the 7-point scale) for the PGIC at end of study (Visit 6 or Early Termination) compared to Visit 1.
Time Frame: End of Randomized treatment period (11 weeks)
Population: All efficacy analyses are based on the Intent-to-Treat population, defined as all randomized patients who received at least one dose of randomized study drug and had at least one post-baseline PGIC assessment.
Measure: Number; unit: participants
Arm/Group | No Treatment Added | Milnacipran Added
Number analyzed (Participants) | 173 | 179
participants
  Responder | 36 | 83
  Non-Responder | 137 | 96
Statistical Analysis 1: Comparison: No Treatment Added vs Milnacipran Added; The responder rates between 'No Treatment Added' and 'Milnacipran Added' groups were compared using a logistic regression model; Test type: Superiority or Other; p < 0.001, Regression, Logistic

2. Secondary Outcome: Change From Baseline in Visual Analog Scale (VAS) 1-week Pain Recall at End of Study
Description: The secondary efficacy measure was the change from Visit 2 (Week 0) in the 1-week pain recall at Visit 6 (Week 11) or End of Study, measured using a 100-mm VAS assessment of pain (0 indicating no pain and 100 indicating the worst possible pain).
Time Frame: Baseline (0 weeks) and End of Randomized Treatment Period (11 weeks)
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | No Treatment Added | Milnacipran Added
Number analyzed (Participants) | 173 | 179
mm | -6.43 (1.93) | -20.77 (1.92)
Statistical Analysis 1: Comparison: No Treatment Added vs Milnacipran Added; This parameter was analyzed using an ANCOVA model with treatment group and study center as factors and baseline value as a covariate; Test type: Superiority or Other; ANCOVA; Least Square Mean Difference = -14.35, 95% CI 2-sided [-18.99 to -9.71]

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events, defined as adverse events which occurred or worsened after starting randomized study drug, were collected from December 2008 to November 2009.
Arm/Group | No Treatment Added | Milnacipran Added
Serious Adverse Events (participants affected / at risk) | 6/178 | 5/184
Other Adverse Events (participants affected / at risk) | 38/178 | 90/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | No Treatment Added (N=178) | Milnacipran Added (N=184)
Suicidal ideation (Psychiatric disorders) | 1 | 2
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Inverteral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Hysterectomy (Surgical and medical procedures) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | No Treatment Added (N=178) | Milnacipran Added (N=184)
Palpitations (Cardiac disorders) | 0 | 10
Nausea (Gastrointestinal disorders) | 5 | 23
Constipation (Gastrointestinal disorders) | 1 | 18
Dry Mouth (Gastrointestinal disorders) | 0 | 10
Fatigue (General disorders) | 4 | 19
Oedema peripheral (General disorders) | 15 | 6
Weight Increased (Investigations) | 15 | 12
Headache (Nervous system disorders) | 4 | 17
Dizziness (Nervous system disorders) | 1 | 14
Anxiety (Psychiatric disorders) | 3 | 12
Insomnia (Psychiatric disorders) | 2 | 10
Hot flush (Vascular disorders) | 0 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other